CLINICAL TRIAL: NCT00256828
Title: A Multicenter, Randomized, Open Label, Clinical Trial Comparing a QD Regimen of Didanosine, Lamivudine and Efavirenz With a Standard BID Regimen of Zidovudine, Lamivudine and Efavirenz in the Starting Treatment of Human Immunodeficiency Virus Infection (GESIDA 39/03)
Brief Title: Once a Day (QD) - Twice a Day (BID) Clinical Trial: Didanosine, Lamivudine and Efavirenz Versus Zidovudine, Lamivudine and Efavirenz in the Starting Treatment of HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Trial Agency of HIV Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GESIDA-3903
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2007-10-16 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infections
Keywords: HIV infection; Highly active antiretroviral therapy; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Didanosine; Lamivudine; efavirenz

INTERVENTIONS:
Drug: didanosine + lamivudine + efavirenz

SUMMARY:
The purpose of this study is to compare the antiviral activity of two treatment groups for HIV chronic infection: a QD regimen of didanosine, lamivudine and efavirenz versus a BID regimen of zidovudine, lamivudine and efavirenz. Both will be administered with food in the starting treatment of human immunodeficiency virus infection at Week 48.

DETAILED DESCRIPTION:
The inhibition of HIV replication mediated by HAART causes an actual immunological reconstitution that has been clinically evidenced as a dramatic reduction in mortality, incidence of opportunistic diseases, hospital admissions and costs associated with healthcare in HIV-infected patients, which has been shown since the year 1996. Unfortunately, the eradication of HIV is not feasible with the therapies available; therefore, treatment of HIV infection is currently approached as a "life-long" strategy. HAART is not free from middle and long-term adverse events.

It must be considered that, until relatively recently, the HAART regimens required taking a high number of tablets several times daily, frequently with diet restrictions, which made compliance difficult and improved the quality of life of the patients. In any case, it must be noted that insufficient compliance with HAART can have harmful consequences for the patient, public health and health resources.

The factors predicting compliance with ART can depend on the patient, the healthcare team and the therapeutic regimen.

As mentioned above, until recent dates, HAART has gathered all factors making compliance difficult: long-term duration, over one drug, over one dose daily and presence of adverse events. Therefore, the adequate compliance is an actual challenge for patients and for the health staff and has been considered, with a good criterion, the weak point of antiretroviral treatment.

For all the above, it can be stated that the ideal HAART regimen would be that with few tablets and that could be taken once daily. The expected advantages of QD regimens could include mainly three: first, they will improve compliance, which will have a highly positive effect on the antiviral efficacy of HAART. On the other hand, QD regimens will enable that HAART is better adapted to the lifestyle of the patient and will have a low interference with working hours, so they will be more convenient and improve quality of life. Finally, it must be noted that QD regimens will enable for monitoring HAART directly, and will allow for a relatively significant group of patients in our setting to follow the treatment with a greater guarantee of success, such as those with problems of drug addiction, lack of social support, mental disease and those admitted to penitentiary centers.

The main disadvantage of QD regimens is the virtual lack of large clinical trials comparing this therapeutic approach to other potent, well-established BID regimens. Therefore, it is very interesting to examine this approach in a randomized clinical trial with an adequate design such as that proposed.

The second problem is the consequences that result of missing a dose since this could entail that for some time - in the 24 hours following the failure - the drug concentrations could decrease enough to stop inhibiting viral replication; this could also promote the emergence of viral strains resistant to the drugs. In principle, the implications of missing a dose depend substantially on the pharmacokinetic properties included in the QD regimen (Cmin, half-life, intracellular concentrations, and the IC50 of the HIV of each patient), so that, the higher the drug half-life and the higher the Cmin/IC50 ratio, the higher the probability that alter missing a dose the Cmin persists above the IC50 of the HIV strain of the patient. Therefore, it is important to select drugs with pharmacokinetic profiles and an antiviral potency enough for QD administration (vide infra).

BID regimen (efavirenz + zidovudine + lamivudine):

In this study, we have chosen as BID regimen that containing NNRTI efavirenz (Sustiva®) and Combivir® which is the commercial combination of the NRTI zidovudine + lamivudine, that will lead patients to take one tablet in the morning and 2 tablets at night. We have chosen this regimen (zidovudine + lamivudine + efavirenz) because it is the starting treatment regimen for HIV chronic infection best studied and considered by many as the gold standard for this indication.

QD regimen (efavirenz + didanosine + lamivudine):

The QD regimen will be made up by didanosine (capsule-CT) + lamivudine + efavirenz, a regimen containing three tablets that must be taken together at night and which is the QD regimen with most experience to date. We have chosen as combination of NRTI didanosine and lamivudine, drugs authorized for QD use with a very good safety profile and no interactions with each other and with efavirenz. The combination of didanosine and lamivudine is highly attractive and is in fact recommended for the starting HAART by various agencies though not at the same level as the combination of zidovudine and lamivudine (which can be only administered BID) just because there are less randomized clinical trials with the former than with the latter combination of NRTI. Therefore, one of the strengths of the study is that it proposes the possibility of assessing the combination of didanosine and lamivudine in a starting HAART regimen.

In this study, the patients allocated to the QD regimen containing didanosine (capsule-CT) + lamivudine + efavirenz will take all tablets together at night with dinner. In principle, this involves a minor deviation from the data sheet of didanosine where it is specified that the drug must be taken fasting.

Didanosine is the second antiretroviral drug marketed and, in the last decade, the presentation and dosage form of this drug have improved remarkably, from bags with buffered powder for twice daily administration, with dispersible tablets with buffer, to the current dosage form which is a gastroresistant capsule (capsule-CT) which allows for administration in once daily doses and that, since it has no buffer, has improved substantially the gastric tolerance to the drug.

The formulations of didanosine as powder or buffered dispersible tablets must be taken fasting for absorption to be optimum, since its administration with food reduces significantly drug absorption and plasma concentrations. However, the effect of food on the absorption of capsules-CT does not cause an unequivocal reduction in drug exposure.

Primary Objective:

* To compare the antiviral activity of the two treatment groups (QD vs BID) at Week 48, based on the percentage of patients with HIV-RNA levels <50 c/ml.

Secondary Objectives:

* To compare the percentage of patients responding to the treatment with HIV-RNA levels < 400 c/ml at Week 48, with the same approach of analysis as for the primary objective.
* To compare the time to therapy failure at Week 48 in both treatment regimens.
* To compare the increase in the CD4 cell levels from baseline to Week 48 in both treatment regiments.
* To compare the impact on the quality of life of both treatment regimens.
* To compare compliance of both treatment regimens.
* To compare the safety and tolerance of both treatment regimens along the 48 weeks of treatment.
* To assess the efficacy of the administration of didanosine together with food.

Randomization Procedure:

The randomization will be centralized and stratified by the baseline viral burden level, being higher or lower than 100,000 cop/ml. The patients giving their written informed consent will be included in the study. To include a patient, the clinical trial agency Gesida will be contacted by phone.

Study Procedures:

HIV-RNA, CD4 and routine labs will be collected at screening, baseline, w1, w4, w12, w24 and w48. Quality of life will be measured with a self-patient report questionnaire (MOS-HIV).

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV infection with plasma RNA viral burden of HIV > 2,000 copies/ml obtained in the month prior to randomization.
* Ages 18 years or older.
* Women with childbearing potential should use an effective contraceptive method.
* The subjects should give their written informed consent.
* The subjects should provide the baseline laboratory values measured during the 4 weeks prior to the start of the study drugs, specified below:

  * serum creatinine < 1.5 times the upper normal limit;
  * total amylase < 1.4 times the upper normal limit;
  * liver enzymes (AST, ALT) < 4 times the upper normal limit.

Exclusion Criteria:

* Previous antiretroviral treatment.
* Suspected (acute) primary HIV infection starting less than six months before.
* Suspected or proven acute hepatitis in the 30 days prior to inclusion in the study. Subjects with chronic hepatitis are eligible provided their liver function enzymes < 4 times the upper normal limit.
* Previous therapy with agents with a significant potential of systemic myelosuppression, neurotoxicity, pancreatotoxicity, liver toxicity or cytotoxicity in the 3 months prior to the start of the study, or expected need for requiring therapy on inclusion, or therapy with methadone or ribavirin/interferons or treatment with neurotoxic drugs or drugs affecting CYP 3A4.
* Patients under methadone program
* Abuse of alcohol or drugs, sufficient, in the investigator's opinion, to prevent an adequate compliance with the study treatment or that could increase the risk of developing pancreatitis or toxic hepatitis.
* Untreatable diarrhea (> 6 loose stools/day for at least 7 consecutive days) within the 30 days prior to inclusion in the study.
* Pregnancy or nursing.
* History of bilateral peripheral neuropathy or signs and symptoms of bilateral peripheral neuropathy > Grade 2 on screening.
* Inability to tolerate oral drugs.
* Any other clinical condition or previous therapy that, in the investigator's opinion, leads the patient to be inadequate for the study or unable to comply with the dosage requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360
Dates: Start 2004-06; Study Completion 2006-11

PRIMARY OUTCOMES:
Percentage of patients with HIV-RNA levels < 50 c/ml (intent-to-treat [ITT])

SECONDARY OUTCOMES:
Percentage of patients with HIV-RNA level < 400 c/ml
Time to therapy failure
CD4 cell count increase from Baseline to Week 48 (w48)
Quality of life changes
Compliance to both treatment regimens
Description of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Juan Berenguer Berenguer, MD, Study Chair — Gregorio Marañón Hospital
Locations (57):
- Spain (57):
  - Hospital Universitario de San Juan de Alicante, Alicante, Alicante
  - Hospital General de Área de Elda, Elda, Alicante
  - Hospital de Orihuela-Vega Baja, San Bartolomé-Orihuela, Orihuela, Alicante
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Santa Creu y Sant Pau, Barcelona, Barcelona
  - Hospital General Vall D'Hebrón, Barcelona, Barcelona
  - Hospital de Mollet, Barcelona, Barcelona
  - Consorcio Sanitario de Mataró, Barcelona, Barcelona
  - Hospital De Vic, Barcelona, Barcelona
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital Sant Llorenc de Viladecans, Viladecans, Barcelona
  - Hospital General Yagüe, Burgos, Burgos
  - Hospital General de Jerez de la Frontera11407, Jerez de la Frontera, Cadiz
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Sierrallana de Torrelavega, Torrelavega, Cantabria
  - Hospital General de Castellón, Castellon, Castellon
  - Hospital Provincial Reina Sofía de Córdoba, Córdoba, Cordoba
  - Hospital Provincial Nuestra Señora de la Montaña-Complejo Hospitalario de Cáceres, Cáceres, Cáceres
  - Hospital Comarcal de la Selva, Blanes, Gerona
  - Hospital de Figueres, Figueras, Gerona
  - Hospital de Palamós, Palamós, Gerona
  - Hospital Clínico Universitario San Cecilio, Granada, Granada
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital General San Jorge, Huesca, Huesca
  - Hospital Ciudad de Jaén, Jaén, Jaen
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Arquitecto Marcide, Ferrol, La Coruña
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Carlos Haya, Málaga, Malaga
  - Hospital Virgen de la Victoria, Málaga, Malaga
  - Hospital Comarcal Axarquía de Vélez, Málaga, Malaga
  - Hospital General Universitario de Murcia, Murcia, Murcia
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital de Covadonga-Central de Asturias, Oviedo, Oviedo
  - Complejo Hospitalario de Pontevedra, Pontevedra, Pontevedra
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Xeral-Cíes de Vigo, Vigo, Pontevedra
  - Hospital General-Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General de Segovia, Segovia, Segovia
  - Hospital General Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital La Fe de Valencia, Valencia, Valencia
  - Hospital Doctor Peset, Valencia, Valencia
  - Hospital del Río Hortega, Valladolid, Valladolid
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Virgen de la Concha, Zamora, Zamora
  - Hospital Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Berenguer J, Gonzalez J, Ribera E, Domingo P, Santos J, Miralles P, Angels Ribas M, Asensi V, Gimeno JL, Perez-Molina JA, Terron JA, Santamaria JM, Pedrol E; GESIDA 3903 Team. Didanosine, lamivudine, and efavirenz versus zidovudine, lamivudine, and efavirenz for the initial treatment of HIV type 1 infection: final analysis (48 weeks) of a prospective, randomized, noninferiority clinical trial, GESIDA 3903. Clin Infect Dis. 2008 Oct 15;47(8):1083-92. doi: 10.1086/592114. PMID 18781872